CLINICAL TRIAL: NCT00246337
Title: A Multicenter, Double-Blind, Placebo and Active-Controlled, Dose-Finding Study of MK0974 in the Treatment of Acute Migraine
Brief Title: A Dose-Finding Study of MK0974 in Acute Migraine (MK0974-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-004; 2005_082
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant; rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- Placebo (Placebo Comparator): Placebo to match assigned treatment arm; one orally-administered dose, plus an optional second dose of active drug, per assigned treatment arm, to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: Comparator: Placebo
- MK0974 25 mg (Experimental): MK0974 25 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 50 mg (Experimental): MK0974 50 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 100 mg (Experimental): MK0974 100 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 200 mg (Experimental): MK0974 200 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 300 mg (Experimental): MK0974 300 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 400 mg (Experimental): MK0974 400 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- MK0974 600 mg (Experimental): MK0974 600 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: MK0974
- Rizatriptan 10 mg (Active Comparator): Rizatriptan 10 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  Interventions: Drug: Rizatriptan

INTERVENTIONS:
Drug: Comparator: Placebo — Placebo to match assigned treatment arm; one orally-administered dose
  Arms: Placebo
Drug: MK0974 — MK0974 25 mg; one orally-administered dose
  Arms: MK0974 25 mg
Drug: MK0974 — MK0974 50 mg; one orally-administered dose
  Arms: MK0974 50 mg
Drug: MK0974 — MK0974 100 mg; one orally-administered dose
  Arms: MK0974 100 mg
Drug: MK0974 — MK0974 200 mg; one orally-administered dose
  Arms: MK0974 200 mg
Drug: MK0974 — MK0974 300 mg; one orally-administered dose
  Arms: MK0974 300 mg
Drug: MK0974 — MK0974 400 mg; one orally-administered dose
  Arms: MK0974 400 mg
Drug: MK0974 — MK0974 600 mg; one orally-administered dose
  Arms: MK0974 600 mg
Drug: Rizatriptan — Rizatriptan 10 mg; one orally-administered dose
  Arms: Rizatriptan 10 mg

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of an MK 0974 for migraine headache and to identify an appropriate dose range for further study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has at least 1 year history of migraine (with or without aura)
* Females of childbearing years must use acceptable contraception throughout trial
* Patient is in general good health based on screening assessment

Exclusion Criteria:

* Patient is pregnant/breast-feeding (or is a female expecting to conceive during the study period)
* Patient has heart disease, uncontrolled hypertension (high blood pressure), uncontrolled diabetes or other significant disease
* Patient has major depression, other pain syndromes that might interfere with study assessments, psychiatric conditions, dementia, or significant neurological disorders (other then migraine)
* Patient has a history of gastric or small intestinal surgery or has a disease that causes malabsorption
* Patient has a history of cancer within the last 5 years

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Ho TW, Mannix LK, Fan X, Assaid C, Furtek C, Jones CJ, Lines CR, Rapoport AM; MK-0974 Protocol 004 study group. Randomized controlled trial of an oral CGRP receptor antagonist, MK-0974, in acute treatment of migraine. Neurology. 2008 Apr 15;70(16):1304-12. doi: 10.1212/01.WNL.0000286940.29755.61. Epub 2007 Oct 3. PMID 17914062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 centers from the United States participated. First Patient treated on 01 December 2005; Last Patient Last Treatment was on 01 May 2006.
Pre-assignment Details: Participants were assessed, using the protocol inclusion and exclusion criteria, at Visit 1, and if eligible were randomized at that same visit.
Period: Overall Study
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Started | 147 | 16 | 18 | 17 | 16 | 54 | 54 | 53 | 45
Completed Period (Initial Dose) | 46 | 4 | 9 | 5 | 8 | 29 | 29 | 27 | 19
Completed Period (Both Doses) | 69 | 10 | 6 | 11 | 4 | 10 | 16 | 13 | 15
Completed | 115 | 14 | 15 | 16 | 12 | 39 | 45 | 40 | 34
Not Completed | 32 | 2 | 3 | 1 | 4 | 15 | 9 | 13 | 11
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Qualifying Event | 8 | 2 | 1 | 1 | 1 | 3 | 3 | 2 | 5
Not completed — Site Terminated | 10 | 0 | 0 | 0 | 0 | 7 | 1 | 6 | 2
Not completed — Abnormal baseline lab values | 7 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 4
Not completed — Overwhelmed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violator | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reported as completing trial in error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo to match assigned treatment arm; one orally-administered dose, plus an optional second dose of active drug, per assigned treatment arm, to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 25 mg: MK0974 25 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 50 mg: MK0974 50 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 100 mg: MK0974 100 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 200 mg: MK0974 200 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 300 mg: MK0974 300 mg; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 400 mg: MK0974 400 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 600 mg: MK0974 600 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- Rizatriptan 10 mg: Rizatriptan 10 mg; one orally-administered dose plus an optional second dose (placebo) to treat a single moderate-to-severe migraine headache.
  The reported number of participants are all patients randomized who received study drug and completed the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg | Total
Number analyzed (Participants) | 115 | 14 | 15 | 16 | 12 | 39 | 45 | 40 | 34 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.6) | 43.0 (10.1) | 41.5 (10.9) | 40.9 (7.5) | 34.3 (11.7) | 40.5 (10.4) | 40.1 (11.9) | 44.5 (12.0) | 40.2 (10.8) | 41.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 11 | 14 | 14 | 9 | 34 | 42 | 36 | 28 | 292
  Male | 11 | 3 | 1 | 2 | 3 | 5 | 3 | 4 | 6 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 92 | 10 | 11 | 11 | 6 | 29 | 34 | 38 | 28 | 259
  Black | 18 | 4 | 3 | 3 | 5 | 7 | 10 | 2 | 5 | 57
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  European | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hispanic American | 4 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 9
  Multi-Racial | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Baseline Severity [Number; unit: Participants] — Baseline severity was self-reported by the participant and recorded in the take-home diary. Migraine pain was rated on a 4-point scale (No Pain=0, Mild Pain=1, Moderate Pain=2, Severe Pain=3).
  Participants
    Moderate | 81 | 11 | 9 | 15 | 6 | 26 | 34 | 30 | 27 | 239
    Severe | 34 | 3 | 6 | 1 | 6 | 12 | 11 | 10 | 7 | 90
    Baseline Severity data missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild), 2 (moderate), 3 (severe). Pain Relief is defined as participants reporting relief from moderate to severe migraine headache (Grade 2 or 3) to mild or none (Grade 1 or 0) in the setting of a typical migraine attack.
Time Frame: 2 hours post dose
Population: All Patients Treated (APT): included all randomized participants who took study medication and reported the post-dose assessment of the primary efficacy measure. Patients were counted in the treatment group to which they were randomized.
  One patient in the MK974 300 mg group was excluded because baseline headache severity information was missing.
Measure: Number; unit: Participants
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 115 | 14 | 15 | 16 | 12 | 38 | 45 | 40 | 34
Participants | 52 | 5 | 9 | 8 | 5 | 25 | 22 | 27 | 24
Statistical Analysis 1: Comparison: Placebo vs MK0974 300 mg vs MK0974 400 mg vs MK0974 600 mg; Only the MK0974 300mg, 400mg, and 600mg groups are included in the comparison with placebo based on the protocol-specified test statistics selection and the fact that all lower doses were discontinued after the interim analysis. Overall power =85%; Test type: Superiority or Other; p = 0.015, generalized linear model — 0.05 is the pre-specified significance level; The p-value is based on the average response of the MK0974 200mg, 400mg, and 600mg groups vs. placebo

2. Secondary Outcome: Pain Freedom at 2 Hours
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild), 2 (moderate), 3 (severe). Pain freedom is defined as no pain (Grade 0) at 2 hours post dose.
Time Frame: 2 hours post dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 115 | 14 | 15 | 16 | 12 | 38 | 45 | 40 | 34
Participants | 16 | 3 | 7 | 3 | 2 | 17 | 11 | 13 | 11
Statistical Analysis 1: Comparison: Placebo vs MK0974 300 mg vs MK0974 400 mg vs MK0974 600 mg; Only the MK0974 300mg, 400mg, and 600mg groups are included in the comparison with placebo based on the protocol-specified test statistics selection and the fact that all lower doses were discontinued after the interim analysis; Test type: Superiority or Other; p < 0.001, generalized linear model — 0.05 is the pre-specified significance level; The p-value is based on the average response of the MK0974 200mg, 400mg, and 600mg groups vs. placebo

3. Secondary Outcome: Sustained Pain Relief
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild), 2 (moderate), 3 (severe). Sustained pain relief is defined as pain relief at 2 hours and no headache recurrence, no need for the optional 2nd dose, or any rescue medication, between 2 and 24 hours post dose.
Time Frame: 2-24 hours post dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 115 | 13 | 15 | 16 | 11 | 38 | 45 | 40 | 34
Participants | 27 | 1 | 9 | 3 | 3 | 20 | 17 | 21 | 12
Statistical Analysis 1: Comparison: Placebo vs MK0974 300 mg vs MK0974 400 mg vs MK0974 600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, generalized linear model — 0.05 is the pre-specified significance level

4. Secondary Outcome: Sustained Pain Freedom
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild), 2 (moderate), 3 (severe). Sustained pain freedom is defined as pain freedom at 2 hours and no headache return to mild/moderate/severe, no need for the optional 2nd dose, or any rescue medication, between 2 and 24 hours post dose.
Time Frame: 2-24 hours post dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 115 | 13 | 15 | 16 | 11 | 38 | 45 | 40 | 34
Participants | 12 | 1 | 7 | 3 | 1 | 15 | 10 | 13 | 6
Statistical Analysis 1: Comparison: Placebo vs MK0974 300 mg vs MK0974 400 mg vs MK0974 600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, generalized linear model — 0.05 is the pre-specified significance level; The p-value is based on the average response of the MK0974 200mg, 400mg, and 600mg groups vs. placebo

ADVERSE EVENTS:
Time Frame: Within 14 Days Post-Dose. The numbers in the Participant Flow reflect all patients randomized.
Description: For safety, the population was based on actual treatment with any dose (first dose, or the optional second dose which they could take after 4 hours). Patients were counted based on actual treatment (including the optional second dose). If the patient was treated with both placebo and active, they were counted under the active treatment group.
Arm/Group | Placebo | MK0974 25 mg | MK0974 50 mg | MK0974 100 mg | MK0974 200 mg | MK0974 300 mg | MK0974 400 mg | MK0974 600 mg | Rizatriptan 10 mg
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/17 | 0/19 | 0/27 | 0/18 | 0/51 | 0/52 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 10/47 | 4/17 | 9/19 | 4/27 | 7/18 | 9/51 | 12/52 | 14/49 | 10/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | MK0974 25 mg (N=17) | MK0974 50 mg (N=19) | MK0974 100 mg (N=27) | MK0974 200 mg (N=18) | MK0974 300 mg (N=51) | MK0974 400 mg (N=52) | MK0974 600 mg (N=49) | Rizatriptan 10 mg (N=50)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | MK0974 25 mg (N=17) | MK0974 50 mg (N=19) | MK0974 100 mg (N=27) | MK0974 200 mg (N=18) | MK0974 300 mg (N=51) | MK0974 400 mg (N=52) | MK0974 600 mg (N=49) | Rizatriptan 10 mg (N=50)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 0 | 0 | 1 | 0 | 3 | 5 | 5 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 0 | 2 | 3 | 1 | 4 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 4 | 2
Bruxism (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.